CLINICAL TRIAL: NCT04891081
Title: Plasma Metanephrines in Patients With Cyanotic and Acyanotic Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Principal Investigator, Mojca Jensterle, Clinical Professor, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0000
Record Dates: First submitted 2021-05-10; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Acyanotic Congenital Heart Disease; Cyanotic Congenital Heart Disease; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cyanotic Congenital Heart Disease
- Patients with acyanotic Congenital Heart Disease

SUMMARY:
The aim of our study is to compare plasma metanephrines in patients with cyanotic and acyanotic congenital heart disease and possible association with chronic hypoxic stress.

ELIGIBILITY:
Inclusion Criteria:

* patients with congenital heart disease attending regular follow up

Exclusion Criteria:

* missing main data in medical documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with congenital heart disease attending regular follow ups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-09 (Estimated)

PRIMARY OUTCOMES:
Plasma metanephrine level | baseline, one point of time in a cross-sectional study
  Level of plasma metanephrine
Plasma normetanephrine level | baseline, one point of time in a cross-sectional study
  Level of plasma normetanephrine

SECONDARY OUTCOMES:
Hypoxemia | baseline, one point of time in a cross-sectional study
  Length of hypoxemia presence in years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, University of Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No